CLINICAL TRIAL: NCT01838200
Title: A Phase I Study of Intralesional Bacillus Calmette-Guerin (BCG) and Followed by Ipilimumab Therapy in Patients With Advanced Metastatic Melanoma
Brief Title: Phase I Study of Intralesional Bacillus Calmette-Guerin (BCG) Followed by Ipilimumab in Advanced Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment due to changes in standard of care
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2012-003
Record Dates: First submitted 2013-04-17; First posted 2013-04-23 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Melanoma
Keywords: BCG; Bacillus Calmette-Guérin; Ipilimumab; YERVOY; Advanced Metastatic Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — BCG Vaccine; Ipilimumab; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) (Experimental): Patients with an induration <10 mm in diameter after the baseline PPD reactivity test received BCG (IL) on Day 1, followed by isoniazid (orally, daily) starting 28 days after the BCG injection and continuing for 4 weeks, and ipilimumab (IV) administered every 3 weeks starting 5 weeks after the BCG injection and continuing for a total of 4 doses.
  Interventions: Biological: Bacillus Calmette-Guérin (BCG) vaccine; Drug: Ipilimumab; Drug: Isoniazid
- Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU) (Experimental): Patients with an induration <10 mm in diameter after the baseline PPD reactivity test received BCG (IL) on Day 1, followed by isoniazid (orally, daily) starting 28 days after the BCG injection and continuing for 4 weeks, and ipilimumab (IV) administered every 3 weeks starting 5 weeks after the BCG injection and continuing for a total of 4 doses.
  Interventions: Biological: Bacillus Calmette-Guérin (BCG) vaccine; Drug: Ipilimumab; Drug: Isoniazid
- Cohort 1, Group 3 (BCG 4.0-16.0 × 10^6 CFU) (Experimental): Patients with an induration <10 mm in diameter after the baseline PPD reactivity test were to receive BCG (IL) on Day 1, followed by isoniazid (orally, daily) starting 28 days after the BCG injection and continuing for 4 weeks, and ipilimumab (IV) administered every 3 weeks starting 5 weeks after the BCG injection and continuing for a total of 4 doses.
  Interventions: Biological: Bacillus Calmette-Guérin (BCG) vaccine; Drug: Ipilimumab; Drug: Isoniazid
- Cohort 2 (BCG 0.16-0.64 × 10^6 CFU) (Experimental): Patients with an induration ≥10 mm in diameter after the baseline PPD reactivity test were to receive BCG (IL) on Day 1, followed by isoniazid (orally, daily) starting 28 days after the BCG injection and continuing for 4 weeks, and ipilimumab (IV) administered every 3 weeks starting 5 weeks after the BCG injection and continuing for a total of 4 doses.
  Interventions: Biological: Bacillus Calmette-Guérin (BCG) vaccine; Drug: Ipilimumab; Drug: Isoniazid

INTERVENTIONS:
Biological: Bacillus Calmette-Guérin (BCG) vaccine — BCG was to be administered as a single intralesional injection (200 µL volume) on Day 1 at varying doses depending on cohort assignment.
  Other Names: BCG
Drug: Ipilimumab — Ipilimumab was to be administered as a 90-minute IV infusion at a dose of 3 mg/kg every 3 weeks (± 3 days) on Days 36, 57, 78, and 99.
  Other Names: YERVOY
Drug: Isoniazid — Isoniazid was to be administered orally at a dose of 300 mg (3 × 100 mg tablets) every day from Days 29 through 56.

SUMMARY:
This was a Phase 1, open-label, dose-escalation, single-center study in patients with histologically confirmed Stage III or IV melanoma and at least 3 metastatic cutaneous or subcutaneous lesions that were suitable and accessible for intralesional (IL) injection (1 lesion), biopsy (1 lesion), and response evaluation (1 lesion). The primary objective was to determine the safety of IL administration of bacillus Calmette-Guerin (BCG) followed by oral dosing with an antibiotic (isoniazid) and intravenous (IV) infusions of ipilimumab. Secondary objectives were to evaluate the clinical efficacy (induction of tumor response) and immunogenicity (induction of immune response against the tumors) of the combination regimen.

DETAILED DESCRIPTION:
Patients were enrolled into one of two study cohorts depending on the induration noted after a baseline purified protein derivative (PPD) skin test to determine tuberculin reactivity. Cohort 1 comprised patients with an induration of <10mm in diameter, and Cohort 2 comprised patients with an induration of ≥10mm. Enrollment was staggered by 3 weeks for each of the first 3 patients in Cohort 1, Group 1 to enable safety monitoring of each patient prior to exposure of additional patients.

In all cohorts, study treatment included BCG (200 µL volume) given IL on Day 1, isoniazid (300 mg) given orally daily from Days 29 to 56, and ipilimumab (3 mg/kg) given IV every 3 weeks (± 3 days) on Days 36, 57, 78, and 99. The dose of BCG varied by assigned treatment group: Cohort 1, Group 1 received 0.16 - 0.64 × 10^6 colony-forming units (CFU); Cohort 1, Group 2 received 0.8 - 3.2 x 10^6 CFU; Cohort 1, Group 3 was to receive 4.0 - 16.0 x 10^6 CFU; and Cohort 2 was to receive 0.16 - 0.64 × 10^6 CFU. Enrollment into Cohort 2 was to be initiated after the final patient in Cohort 1, Group 1 reached Week 7. Enrollment was then to proceed in parallel for Cohort 2 and Cohort 1, Groups 2 and 3.

Patients were monitored for safety, tumor response, and immunogenicity (cellular, humoral, and in situ immunity) for the duration of study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage III (unresectable) or stage IV melanoma.
2. Minimum 1 metastatic lesion, cutaneous or subcutaneous, but ideally 3 or more lesions, to accommodate intralesional injection (1 lesion), accessibility for biopsy (1 lesion), and evaluability for response by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (1 lesion) and modified RECIST (immune-related response criteria [irRC]).
3. Performance status of Eastern Cooperative Oncology Group 0-1.
4. Within the last 2 weeks prior to study Day 1, vital laboratory parameters must have been within normal ranges, except for the following laboratory parameters, which must have been within the ranges specified:

   * Hemoglobin: ≥ 100 g/L
   * Platelets: ≥ 100 x 10^9/L
   * International normalized ratio: ≤ 2.0
   * Creatinine: ≤ 120 µmol/L
   * Bilirubin: ≤ 30 µmol/L
   * Estimated glomerular filtration rate: > 0.75 x lower limit of normal
   * Aspartate and alanine aminotransferase: ≤ 2.0 x upper limit of normal
   * Albumin: > 28 g/L
   * Neutrophils: > 1.5 x 10^9/L
   * Lymphocytes: > 0.5 x 10^9/L
5. Estimated life expectancy of at least 4 to 6 months. Because of the slow onset of action of ipilimumab and the protocol requirement for a 5-week delay post-BCG, patients with rapidly progressive disease may not have been suitable for the protocol.
6. Full recovery from surgery. A minimum of 2 weeks should have elapsed since the most recent surgery.
7. Men and women ≥ 18 years of age.
8. Able and willing to give written informed consent.

Exclusion Criteria:

1. Active cerebral metastases unless stable after radiation for at least 1 month and not requiring corticosteroid treatment for 30 days prior to enrollment.
2. Other known malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
3. History of tuberculosis.
4. History of hypersensitivity to BCG.
5. Any contraindication to the use of isoniazid.
6. Generalized skin disease.
7. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, were excluded from this study, as were patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis). Exceptions: vitiligo, type I diabetes, pernicious anemia (treated).
8. Any underlying medical or psychiatric condition, which in the opinion of the Investigator would have made the administration of ipilimumab hazardous or obscured the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea.
9. Prior immunotherapy or systemic adjuvant therapy for melanoma following most recent relapse and/or resection of melanoma.
10. Prior treatment with a cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) inhibitor.
11. Concomitant therapy with any of the following: interleukin 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids.
12. Known human immunodeficiency virus positivity, Hepatitis B or Hepatitis C.
13. Chemotherapy or radiation therapy within the preceding 4 weeks (6 weeks for nitrosourea drugs).
14. Lack of availability for immunological and clinical follow-up assessments.
15. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing.
16. Mental impairment that may have compromised the ability to give informed consent and to comply with the requirements of the study.
17. Women who were pregnant (positive pregnancy test at baseline), or breastfeeding.
18. Men and women unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug.
19. Prisoners or patients who were compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-08-17 (Actual); Study Completion 2015-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cebon, MD, PhD, Principal Investigator — Austin Health
Locations (1):
- Austin Health, LICR Melbourne Austin Branch, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Da Gama Duarte J, Parakh S, Andrews MC, Woods K, Pasam A, Tutuka C, Ostrouska S, Blackburn JM, Behren A, Cebon J. Autoantibodies May Predict Immune-Related Toxicity: Results from a Phase I Study of Intralesional Bacillus Calmette-Guerin followed by Ipilimumab in Patients with Advanced Metastatic Melanoma. Front Immunol. 2018 Mar 2;9:411. doi: 10.3389/fimmu.2018.00411. eCollection 2018. PMID 29552014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early due to slow enrollment; thus, Cohort 1 Group 3 and Cohort 2 were not enrolled.
Groups:
- Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU): Patients with an induration <10 mm in diameter after the baseline PPD reactivity test received BCG (IL, 200 µL volume) at a dose of 0.16 - 0.64 × 10^6 CFU on Day 1. Isoniazid (300 mg) was administered orally every day from Days 29 through 56. Ipilimumab (3 mg/kg) was administered as a 90-minute IV infusion every 3 weeks (± 3 days) on Days 36, 57, 78, and 99.
- Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU): Patients with an induration <10 mm in diameter after the baseline PPD reactivity test received BCG (IL, 200 µL volume) at a dose of 0.8 - 3.2 × 10^6 CFU on Day 1. Isoniazid (300 mg) was administered orally every day from Days 29 through 56. Ipilimumab (3 mg/kg) was administered as a 90-minute IV infusion every 3 weeks (± 3 days) on Days 36, 57, 78, and 99.
Period: Overall Study
Arm/Group | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU)
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Progressive disease | 3 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 61.3 [50 to 70] | 53.5 [43 to 64] | 58.2 [43 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 2 | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    0 | 2 | 0 | 2
    1 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period. Dose-limiting toxicity (DLT) for BCG was defined as any ≥ Grade 3 local injection site reaction (ulceration or necrosis requiring operative intervention), and DLT for ipilimumab was defined as any toxicity that required dosing modifications in accordance with the recommendations in the local product labelling, or any ≥ Grade 3 hematologic or nonhematologic toxicity that was definitely, probably, or possibly related to the administration of ipilimumab.
Time Frame: Continuously for up to 5 months
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU)
Number analyzed (Participants) | 3 | 2
Participants
  Any TEAE | 3 | 2
  Maximum grade 1 TEAE | 0 | 0
  Maximum grade 2 TEAE | 1 | 0
  Maximum grade 3 TEAE | 2 | 1
  Maximum grade 4 TEAE | 0 | 1
  BCG-related TEAE | 0 | 1
  Ipilimumab-related TEAE | 1 | 2
  Isoniazid-related TEAE | 0 | 0
  Serious TEAE | 2 | 1
  TEAE Leading to BCG Discontinuation | 0 | 0
  TEAE Leading to Ipilimumab Discontinuation | 1 | 2
  TEAE Leading to Isoniazid Discontinuation | 0 | 0
  TEAE Meeting DLT Criteria | 0 | 2

2. Secondary Outcome: Number of Patients With Best Overall Clinical Tumor Response
Description: Tumor responses were evaluated using computed tomography and clinical photography at Baseline, Weeks 6, 17, 21, and 30 (± 3-day window for each assessment), and at the end of the study. Tumor response was designated according to the Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1). Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions (no evaluable disease); Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 5 months
Population: The Efficacy Analysis Set includes all patients who received at least 1 dose of study treatment and had response evaluated through Week 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU)
Number analyzed (Participants) | 3 | 2
Participants
  Best response: SD | 2 | 0
  Best response: PD | 1 | 2

3. Secondary Outcome: Number of Patients With Best Overall Immune-related Tumor Response
Description: Immune-related tumor responses were evaluated using computed tomography and clinical photography at Baseline, Weeks 6, 17, 21, and 30 (± 3-day window for each assessment), and at the end of the study. Tumor response was designated according to the immune-related Response Criteria (irRC) (Wolchok et al. Clin Cancer Res 2009;15:7412-20) into the following categories: immune-related complete response (irCR) requires disappearance of all lesions in two consecutive observations not less than 4 weeks apart; immune-related partial response (irPR) requires ≥ 50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart; immune-related stable disease (irSD) is assigned when neither a 50% decrease from baseline tumor burden nor a 25% increase in tumor burden from nadir can be established; immune-related progressive disease (irPD) requires a ≥ 25% increase from nadir in tumor burden at any single time point in two consecutive observations at least 4 weeks apart.
Time Frame: Up to 5 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU)
Number analyzed (Participants) | 3 | 2
Participants
  Best response: irSD | 1 | 1
  Best response: irPD | 2 | 0
  Not evaluable by irRC | 0 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs) and are presented in the summary tabulations. The AE reporting period for this study was up to 5 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.0), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) (N=3) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU) (N=2)
Colitis (Gastrointestinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Group 1 (BCG 0.16-0.64 × 10^6 CFU) (N=3) | Cohort 1, Group 2 (BCG 0.8-3.2 × 10^6 CFU) (N=2)
Fatigue (General disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Axillary pain (General disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Influenza-like illness (General disorders) | 1 | 0
Injection site ulcer (General disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As the study was terminated early due to slow enrollment, immune response (cellular, humoral, in situ) analyses were not performed as outlined in the protocol due to small sample sizes within each arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less